CLINICAL TRIAL: NCT00706927
Title: A Double-masked Randomized Cross-over Study Comparing of the Effect of Xalacom® (Latanoprost/Timolol)and Combigan® (Brimonidine/Timolol) Fixed Combination on Intraocular Pressure and Ocular Blood Flow in Patients With Primary Open Angle Glaucoma or Ocular Hypertension
Brief Title: Effect of Xalacom® (Latanoprost/Timolol) and Combigan® (Brimonidine/Timolol) Fixed Combination on Intraocular Pressure and Ocular Blood Flow in Patients With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. - Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPHT-241005
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Retina; Ocular Physiology
Keywords: xalacom; combigan; ocular blood flow
MeSH Terms: interventions — Latanoprost; Xalacom; Timolol; Brimonidine Tartrate, Timolol Maleate Drug Combination; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: latanoprost 0.005% + timolol 0,5% fixed combination — 1 drop per day and eye for 6 weeks
  Other Names: Xalacom® (latanoprost/timolol)
Drug: brimonidine 0,2% + timolol 0,5% fixed combination — 1 drop twice a day per eye for 6 weeks
  Other Names: Combigan® (brimonidine/timolol)

SUMMARY:
Glaucoma is one of the most common causes of blindness in the industrialized nations. For a long time glaucoma has been defined as a disease in which high intraocular pressure (IOP) leads to irreversible optic disc damage and subsequent visual field loss. However, recent investigations show that IOP is not the only factor that is involved in the glaucomatous process leading to retinal ganglion cell death. The role of vascular factors in the pathogenesis of glaucoma has recently received much attention based on animal experiments and epidemiological studies. The main focus of glaucoma is still directed towards a decrease in IOP. There is, however, also considerable interest whether antiglaucoma drugs influence ocular perfusion. Although measurement of ocular blood flow is still difficult, a number of innovative techniques have been realized which cover different aspects of ocular perfusion. In the present study Xalacom® (latanoprost/timolol) and the fixed combination of Combigan® (brimonidine/timolol) will be compared with respect to their IOP lowering efficacy as well as their ocular hemodynamic effects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years
* Unilateral or bilateral primary open angle glaucoma, ocular hypertension, exfoliation glaucoma, pigmentary glaucoma with IOP between 22 -35mmHg
* At least 3 reliable visual field testings
* 4 weeks for ß adrenergic receptor antagonists and prostaglandin analogues, 2 weeks for adrenergic agonists, and 5 days for cholinergic agonists and carbonic anhydrase inhibitors

Exclusion Criteria:

* History of acute angle closure
* Closed or barely open anterior chamber angle
* Mean deviation of visual field testing > 10
* Intraocular surgery or argon laser trabeculoplasty within the last six months
* Ocular inflammation or infection within the last three months
* Contact lenses
* Patients with bradycardia (heart rate < 50 beats/min)
* Second and third degree heart block
* Asthma
* COPD
* Congestive heart failure
* Severe renal impairment (creatinine clearance < 1.8 L/h)
* History of hypersensitivity to one of the study drugs or drugs with similar chemical structure
* Topical or systematically/oral therapy with steroids
* History of non-IOP responder to beta-blockers, alpha-2 adrenergic or prostaglandin analogues
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-01; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Optic disc blood flow measured with laser Doppler flowmeter (rel units) | 12 weeks
Intraocular pressure (mmHg) | 12 weeks

SECONDARY OUTCOMES:
Retrobulbar flow velocities as measured with color Doppler imaging (cm/s) | 12 weeks
Mean defect of visual field measured with automated perimetry (dB) | 12 weeks
Corneal thickness as measured with pachymetry (µm) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria